CLINICAL TRIAL: NCT04171973
Title: Evaluation of Electric Wheelchair Driving Performance in Simulator Compared to Driving in a Real-life Situation, in a Population of Regular Drivers With Neurological Disorders
Brief Title: Evaluation of Electric Wheelchair Driving Performance in Simulator Compared to Driving in Real-life Situations
Acronym: SIMADAPT1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pôle Saint Hélier (Other)
Collaborators: INSA Rennes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2019-A01903-54
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2019-11

CONDITIONS: Neurologic Disorder
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: It is a pilot, prospective, monocentric, controlled, randomized, open-arms, open-ended, minimal risk and minimal constraint study (RIPH category 2).
Masking Description: Neither patients nor evaluators can be unaware of which group they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Driving an electric wheelchair in real condition (Other): In order to be able to evaluate the feasibility of virtual reality driving training, the driving performance will be evaluated on the same 3 standardized circuits: for the control group, 3 circuits of test of pipes in real condition of increasing difficulty are tested. Patients perform 2 passes in this condition.
  Interventions: Device: Driving an electric wheelchair in real condition
- Driving an electric wheelchair in virtual condition (Experimental): In order to be able to evaluate the feasibility of driving training in virtual reality, the driving performance will be evaluated on the same 3 standardized circuits: for the virtual reality group, the circuits have been digitized. Patients perform 2 passes in this condition.
  Interventions: Device: Driving an electric wheelchair in virtual condition

INTERVENTIONS:
Device: Driving an electric wheelchair in real condition — For the control group, 3 test circuits of pipes in real condition of increasing difficulty are tested. Patients perform 2 passes in this condition.
  Arms: Driving an electric wheelchair in real condition
Device: Driving an electric wheelchair in virtual condition — For the virtual reality group, the circuits have been digitized. Patients perform 2 passes in this condition.
  Arms: Driving an electric wheelchair in virtual condition

SUMMARY:
The device that is the subject of this investigation is a solution for driving simulation of an electric wheelchair. It is intended to enable patients who are likely to acquire an electric wheelchair to train in a virtual environment, favorable to the safety of training, to its repetition, and to produce more varied, rich training environments and more tailored to specific and individualized needs. These solutions will make it easier to access real-world driving for patients who are currently experiencing learning difficulties.

It is expected that this investigation demonstrates the reproducibility of driving performance in electric wheelchair driving simulator compared to the real world.

DETAILED DESCRIPTION:
As part of this investigation, it is expected to develop a driving simulator that could contribute to improving the learning of electric wheelchair driving and access to electric wheelchair for people who can not currently claim for physical risks and weak psychology for the participant in the research.

The present clinical investigation aims at evaluating the performances, the safety and the satisfaction of the users with regard to a simulator of driving of electric wheelchair in virtual reality.

The main objective is to evaluate the feasibility of a virtual electric wheelchair driving training, comparing driving performance in virtual reality versus reality, in identical real and virtual standardized circuits, in regular users of electric wheelchairs with neurological disorders.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, over 18 years old,
* Having freely consented to participate in the study,
* With neurological degenerative disorders including cerebrovascular accident and head trauma or neurodegeneration including Parkinson's disease and related syndromes, multiple sclerosis, myopathy and amyotrophic lateral sclerosis,
* Having benefited from an electric wheelchair prescription and traveling in electric wheelchair for more than 3 months,
* Whose electric wheelchair is the main mode of travel,
* The physical measurements (weight, size) are compatible with the use of the physical simulator chosen for the development of the robotic assistance module, according to manufacturer's data 140 kg max and 51 cm max of seat width .

Exclusion Criteria:

* Understanding difficulties preventing the realization of the protocol,
* Motor disorders of the upper limb requiring additional driving technical assistance,
* Patient having expressed difficulties impacting his safety of sedan and / or external, objectified by a negative answer to more than one item on the self-questionnaire WST QF for the items pertaining to driving (6 to 12 and 17 to 28):

  1. inability to perform certain driving tasks (answer "no")
  2. or insecure to achieve them (answer "not at all").
* pregnant, parturient or nursing mother,
* Person deprived of liberty by a judicial or administrative decision, persons under psychiatric care or admitted to a health or social institution for purposes other than research,
* Minor,
* Major under legal protection or unable to express his consent,
* Person in emergency situation who can not express their prior consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-01-29 (Actual)

PRIMARY OUTCOMES:
Number of collision | Day 1
  The primary judgment criterion is the number of collisions on different standardized circuits in real condition versus virtual condition
Number of collision | Day 8
  The primary judgment criterion is the number of collisions on different standardized circuits in real condition versus virtual condition
Number of collision | Day 15
  The primary judgment criterion is the number of collisions on different standardized circuits in real condition versus virtual condition

SECONDARY OUTCOMES:
Driving Speed | Day 1, Day 8 and Day 15
  Speed measured by the completion time of the course on the different circuits in real condition versus virtual condition
Wheelchair Skill Test (WST) | Day 1, Day 8 and Day 15
  Driving performance measured by the Wheelchair Skill Test items corresponding to the different courses in real condition versus virtual condition
NASA-Task Load Index | Day 1, Day 8 and Day 15
  The cognitive load of tests under both conditions will be measured by the NASA-Task Load Index. It is in the form of six scales where the participant must assign a score between zero and one hundred to each of them, score indicating a growing level of intensity. Three dimensions relate to the demands imposed on the subject (mental, physical and temporal demands) and three to the interaction of a subject with the task (effort, frustration and performance)
Ease of Use Questionnaire | Day 1, Day 8 and Day 15
  The satisfaction of the use of the electric wheelchair under the conditions will be evaluated by the self-questionnaire Ease of Use Questionnaire. It measures the subjective usability of a product or service. It is a 30-item survey that examines four dimensions of usability: usefulness, ease of use, ease of learning, and satisfaction. The questionnaires were constructed as seven-point Likert rating scales. Users were asked to rate agreement with the statements, ranging from strongly disagree (1) to strongly agree (7).
Unified theory of acceptance of technology questionnaire (UTAUT) | Day 1, Day 8 and Day 15
  Questionnaire of acceptability / acceptance of the tool and its use by patients based on the Unified Theory of Acceptance and Use Technology (UTAUT).
Igroup Presence Questionnaire (IPQ) | Day 1, Day 8 and Day 15
  The IPQ comprises 14 items rated on a seven-point Likert Scale ranging from -3 to 3. The general item assesses the general "sense of being there", and has high loadings on all three factors, with an especially strong loading on Spatial Presence. The Spatial Presence sub-scale is related to the sense of being physically inside the virtual environment. The involvement sub-scale is directed to evaluate the attention devoted to the virtual environment. The realness sub-scale evaluates the sense of reality attributed to the virtual environment.
The learning effect | Day 1, Day 8 and Day 15
  The learning effect on the virtual circuit and on the real circuit, will be evaluated by progression / stabilization of the time of realization during the sequence of repetitions.
Graybiel score | Day 1, Day 8 and Day 15
  Assessment of discomfort and motion sickness to quantify the intensity of different symptoms during motion sickness.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Gallien, Doctor, Principal Investigator — Pôle Saint Hélier
Locations (1):
- Pole Saint-Hélier, Rennes, Brittany Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fraudet B, Leblong E, Piette P, Nicolas B, Gouranton V, Babel M, Devigne L, Pasteau F, Gallien P. Evaluation of power wheelchair driving performance in simulator compared to driving in real-life situations: the SIMADAPT (simulator ADAPT) project-a pilot study. J Neuroeng Rehabil. 2024 Apr 23;21(1):60. doi: 10.1186/s12984-024-01354-5. PMID 38654367